CLINICAL TRIAL: NCT06679270
Title: An Open-label Extension of APG-20 Study to Evaluate the Long-term Safety and Efficacy of Daily Subcutaneous Metreleptin Treatment in Subjects With Partial Lipodystrophy
Brief Title: Open-label Extension Study to Evaluate Metreleptin in Patients With Partial Lipodystrophy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-20-OLE; APG-20 OLE (Other: Amryt Pharmaceuticals DAC)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Familial Partial Lipodystrophy
Keywords: Metreleptin; familial partial lipodystrophy
MeSH Terms: conditions — Lipodystrophy, Familial Partial | interventions — metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metreleptin (Experimental): Metreleptin [Recombinant-methionyl human Leptin; r-metHuLeptin] for daily injection is a sterile, white, solid lyophilised cake
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Metreleptin is a recombinant human leptin analog that is indicated as an adjunct to diet as replacement therapy to treat the complications of leptin deficiency

SUMMARY:
This Phase 3 study is an Open Label Extension of the APG-20 Study To Evaluate the Long-term Safety and Efficacy of Daily Subcutaneous Metreleptin Treatment in Subjects with Partial Lipodystrophy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥13 years of age, inclusive, at the time of signing the informed consent form (ICF).
2. Subjects must have completed the Parent study APG-20 and, in the opinion of the Investigator and Sponsor, have been compliant with study procedures through Parent study Month 12 visit.
3. Negative pregnancy test (urine or serum) for female subjects of childbearing potential
4. Female subjects must be postmenopausal (defined as cessation of menses for at least 1 year), surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation), or willing to use a highly effective method of contraception (such methods include combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation: oral/intravaginal; transdermal/progestogen-only hormonal contraception associated with inhibition of ovulation: oral/injectable; implantable/intrauterine device [IUD]/intrauterine hormone-releasing system [IUS]/bilateral tubal occlusion/vasectomized partner/sexual abstinence) for the duration of the study (from the time they sign an ICF, until 4 weeks after the last dose of study treatment). Hormonal contraception alone (including oral, injectable, transdermal, and implantable) is not acceptable; an additional barrier method must be used. Intravaginal hormonal contraception or IUS alone are allowed per Investigator's discretion. Subjects on oral contraceptives will not be required to discontinue medication. Subjects will not be permitted to commence oral contraceptives while taking study treatment during the study.
5. Male subjects must be surgically sterile or willing to use an acceptable method of contraception for the duration of the study (from the time they sign an ICF), until 4 weeks after the last dose of study treatment. An acceptable method of contraception would be a barrier method, such as condoms, restraining from having sex, or a partner using the approved methods of contraception for female subjects as per Inclusion Criteria #4.
6. Subjects who are blood/egg/sperm donors should be willing to halt donations during the study and for 4 weeks following their last dose of study treatment.
7. Subjects who are willing to provide informed consent/assent prior to any study-specific procedures. If a minor, the subject has a parent or legal guardian able to read, understand, and sign the ICF and/or a Child Assent Form (if applicable), communicate with the Investigator, and understand and comply with the protocol requirements. Adolescent subjects must also read and understand the Child Assent Form.
8. Subjects who are willing to follow the dietary restrictions recommended by the Investigator.

Exclusion Criteria:

1. Severe hypersensitivity reactions to the study treatment of the Parent study APG-20.
2. Known to have tested positive for human immunodeficiency virus (HIV) or known to be diagnosed with HIV-related LD. Positive HIV test in countries requiring HIV testing.
3. Are immunocompromised or receiving immunomodulatory drugs.
4. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) for subjects ≥18 years of age and by Bedside Schwartz for subjects <18 years of age.
5. Diagnosis of clinically significant hematological abnormalities (including but not limited to clinically significant leukopenia, neutropenia, bone marrow abnormalities, leukemia or lymphoma, or clinically significant pathological lymphadenopathy).
6. Malignancy that is ongoing/not in remission or that currently requires or has required active treatment within the past year (with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ [e.g., breast carcinoma, cervical cancer in situ] that have undergone potentially curative therapy).
7. For females only: currently pregnant (confirmed with a positive pregnancy test) or breastfeeding.
8. Any condition where, in the opinion of the Investigator, participation in this study may pose a significant risk to the subject.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Incidence and Frequency of Treatment-Emergent Adverse Events (Safety and Tolerability) | From enrollment to the end of treatment (until the last participant completes 24 months)
  Incidence and frequency of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs), treatment-related TEAEs, adverse events of special interest (AESI), and adverse events leading to study treatment discontinuation/withdrawal from the study

SECONDARY OUTCOMES:
To evaluate the long-term efficacy (HbA1c) of daily SC metreleptin treatment in participants with familial partial lipodystrophy (FPLD) | From enrollment to the end of treatment (until the last participant completes 24 months)
  Glycated hemoglobin (HbA1c) in participants with HbA1c ≥7% at the Parent study Baseline, over time during the OLE
To evaluate the long-term efficacy (TGs) of daily SC metreleptin treatment in participants with FPLD | From enrollment to the end of treatment (until the last participant completes 24 months)
  - Fasting triglycerides (TGs) in participants with TG ≥500 mg/dL at the Parent study Baseline, over time during the OLE
To evaluate the long-term efficacy (FBG) of daily SC metreleptin treatment in participants with FPLD | From enrollment to the end of treatment (until the last participant completes 24 months)
  * Fasting blood glucose (FBG) in participants with HbA1c ≥7% at the Parent study Baseline, over time during the OLE
  * FBG in participants with FBG above upper limit of normal (ULN) at the Parent study Baseline, over time during the OLE

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Flourish Research, Boca Raton, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbour, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No